CLINICAL TRIAL: NCT00108901
Title: Exercise Dose and Insulin Sensitivity in Obese Children
Brief Title: The Medical College of Georgia PLAY Project: Exercise Dose and Insulin Sensitivity in Obese Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Catherine L. Davis PhD, Principal Investigator, Assoc. Prof. of Pediatrics, Medical College of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60692 (completed); R01DK060692 (NIH); R01DK070922 (NIH)
Record Dates: First submitted 2005-04-20; First posted 2005-04-21 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Type 2 Diabetes Prevention; Executive Function (Cognition)
Keywords: prevention; children; diabetes; overweight; obesity; metabolic syndrome; exercise; insulin resistance; female; male; black, African-American; white, Caucasian; cognition; executive function
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Overweight; Metabolic Syndrome; Motor Activity; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Children were not provided with an after-school exercise intervention. They were free to do their usual activities. Families were offered a monthly healthy lifestyle class.
- Low Dose (Experimental): This group was assigned to receive a 20 min/day aerobic exercise program offered 5 days/week after school. Families were offered a monthly healthy lifestyle class.
  Interventions: Behavioral: Aerobic exercise program
- High dose (Experimental): This group was assigned to receive a 40 min/day aerobic exercise program offered 5 days/week after school. Families were offered a monthly healthy lifestyle class.
  Interventions: Behavioral: Aerobic exercise program

INTERVENTIONS:
Behavioral: Aerobic exercise program — Vigorous intermittent physical activity in group format conducted in research gymnasium after school by research staff. Heart rate monitors documented each child's average heart rate on a daily basis. Small incentives were offered for achieving goal of >150 bpm average HR each day and attending at least 80% of sessions (4 days/week).
  Arms: High dose; Low Dose

SUMMARY:
The study is a behavioral clinical trial of aerobic exercise to determine dose-response effects on risk for type 2 diabetes, fatness, fitness, blood cholesterol levels, and other cardiovascular risk factors in overweight elementary schoolchildren.

The hypothesis is that the more exercise a child does, the more benefit he or she will gain in reducing the risk of diabetes and other cardiovascular diseases.

An ancillary study examined effects on cognition and achievement.

DETAILED DESCRIPTION:
The study is a behavioral clinical trial of aerobic exercise to determine dose-response effects on insulin response to the oral glucose tolerance test, body composition, fitness, lipid profile, inflammation and other metabolic syndrome components in overweight elementary schoolchildren.

Blinded psychological assessments of cognition and achievement were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Overweight, sedentary children
* Black or white race
* Attending specific schools in Augusta, GA area from which this study is recruiting

Exclusion Criteria:

* Unable to participate in testing or vigorous exercise program
* Diabetes
* Taking medication that would affect study results
* Sibling enrolled in project

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2003-06; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Insulin area under the curve (oral glucose tolerance test) | 10-15 weeks
Body composition (% body fat, visceral fat) | 10-15 weeks
Aerobic fitness | 10-15 weeks
Cognition (Executive function) | 10-15 weeks

SECONDARY OUTCOMES:
Glucose (oral glucose tolerance test) | 10-15 weeks
Lipid profile | 10-15 weeks
Inflammation (C-reactive protein, fibrinogen) | 10-15 weeks
Blood pressure | 10-15 weeks
Academic achievement | 10-15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Davis, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Result] Davis CL, Tkacz J, Gregoski M, Boyle CA, Lovrekovic G. Aerobic exercise and snoring in overweight children: a randomized controlled trial. Obesity (Silver Spring). 2006 Nov;14(11):1985-91. doi: 10.1038/oby.2006.232. PMID 17135615
- [Result] Davis CL, Tomporowski PD, Boyle CA, Waller JL, Miller PH, Naglieri JA, Gregoski M. Effects of aerobic exercise on overweight children's cognitive functioning: a randomized controlled trial. Res Q Exerc Sport. 2007 Dec;78(5):510-9. doi: 10.1080/02701367.2007.10599450. PMID 18274222
- [Result] Tomporowski PD, Davis CL, Miller PH, Naglieri JA. Exercise and Children's Intelligence, Cognition, and Academic Achievement. Educ Psychol Rev. 2008 Jun 1;20(2):111-131. doi: 10.1007/s10648-007-9057-0. PMID 19777141
- [Derived] Davis CL, Pollock NK, Waller JL, Allison JD, Dennis BA, Bassali R, Melendez A, Boyle CA, Gower BA. Exercise dose and diabetes risk in overweight and obese children: a randomized controlled trial. JAMA. 2012 Sep 19;308(11):1103-12. doi: 10.1001/2012.jama.10762. PMID 22990269